CLINICAL TRIAL: NCT04025190
Title: Assessing the Feasibility of Screening and Treating Anxiety and Depression in the Bone Marrow Transplant Population
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1704
Record Dates: First submitted 2019-05-07; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Anxiety; Depression
Keywords: anxiety; depression; collaborative care; psycho-oncology; bone marrow transplant
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allogeneic Transplant: All patients seen in the UNC Bone Marrow Transplant clinic who are candidates for allogeneic transplantation attending their pre-admission visit were approached to offer study participation. Study participation included completion of surveys over a time period up to 60 days after their transplant.

SUMMARY:
The primary purpose of this study is twofold: (1) to assess the feasibility of screening adult hematopoietic stem cell transplantation (HSCT) candidates for psychiatric comorbidity (depression and anxiety), and (2) to assess the feasibility of treating depression and anxiety in adult HSCT candidates through a collaborative care algorithm. The ultimate goal of this project is improving HSCT outcomes for allogeneic HSCT candidates by improving identification and treatment of depression and anxiety disorders.

DETAILED DESCRIPTION:
Enrollment and depression and anxiety symptom screening:

All patients who are candidates for allogeneic transplantation and have a scheduled "Pre-Admission Visit" at UNC will be screened by study team to assess if they are eligible for participation. At their "Pre-Admission Visit" patients will be approached for enrollment in the study. Patients who provide written informed consent will complete the Hospital Anxiety and Depression Scale (HADS) survey at that time. If patients screen positive on the HADS (meaning a score of 8 or greater in the anxiety or the depression sections), they will be offered treatment within a collaborative care model intervention. If patients score less than 8 on the HADS survey (negative for symptoms of anxiety or depression) at the Pre-Admission Visit, they will not be offered treatment on study. Their medical records will still be abstracted periodically to follow post-transplant outcomes.

The Collaborative Care Model:

The collaborative care model is a team-delivered treatment program and will be provided by a treatment team of HSCT advanced practice providers (APP), HSCT physician, Comprehensive Cancer Support Program (CCSP) clinicians, and a psychiatrist. The collaborative care treatment intervention will be offered if patients score positive (score of 8 or greater) on the HADS. The collaborative care intervention includes medication consideration, therapy evaluation, and referral to psychiatry if needed.

Treatment Options in the Collaborative Care Model:

There will be three treatment options in the collaborative care model that will be offered to patients who score 8 or greater on the HADS - pharmacologic therapy, non-pharmacologic therapy, or both. If a patient chooses to start pharmacologic therapy after discussion with the APP at the Pre-Admission Visit, this treatment will include one of two antidepressants, which are standard-of-care treatments in medicine. The nonpharmacologic treatment in the Collaborative Care Model will involve a therapy consultation by the CCSP once patient is admitted to the hospital for their HSCT. Patients can also opt to take part in therapy with CCSP as well as taking medications.

The study team at the time of enrollment will gather patient demographics and clinical information including gender, age, disease type, donor HLA match, and history of mental health disorders from the medical record.

Follow-up HADS Surveys:

On Day 0, (day of stem cell infusion) to the hospital for HSCT, patients will undergo another HADS survey, and this will be repeated at Day +14 (+/- 3 days), Day +30 (+/- 3 days), and Day +60 (+/- 3 days). Information will be gathered from the medical records on Day +14, Day +30, and Day +60 regarding symptoms of mucositis, inability to tolerate oral medications, development of hospital-acquired illnesses, ICU admissions, reactivation of viruses (i.e. CMV), readmission to hospital, engraftment status, development of GVHD, and missed clinic appointments.

During the course of the study, all cases will be reviewed weekly in meetings with the psychiatrist and HSCT APPs to address mood symptoms, evaluate the need for titration of medications, and evaluate the need for psychotherapy, provided by CCSP therapist or psychiatrist.

Satisfaction Surveys:

At six months from initial patient enrollment, satisfaction surveys will be distributed to the HSCT APPs and HSCT physicians who have taken part in the study. Each patient at the end of study will also complete a satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* hematological or non-hematological malignancy
* plan to receive an allogeneic stem cell transplant
* patient at UNC's ambulatory BMT clinic
* able to complete self-report measures
* English speaking

Exclusion Criteria:

* plan to receive an autologous transplant
* plan to receive allogeneic transplant for a non-malignancy
* unable to complete self report measures in English
* pregnant
* pre-existing diagnoses of bipolar affective disorder, schizoaffective disorder or schizophrenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients were English speaking adults (age >18 years) with hematological or non-hematological malignancy with an indication to undergo allogeneic HSCT, who were scheduled to undergo allogeneic transplant within 30 days of enrollment, had a scheduled Pre-Transplant Admission clinic visit at the ambulatory HSCT clinic, and were able to complete self-report measures. Patients were excluded if they were pregnant, unable to complete self-report measures in English, or had pre-existing diagnoses of bipolar affective disorder, schizoaffective disorder or schizophrenia.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Systematic screening for depression and anxiety using the Hospital Anxiety and Depression Scale | Day 0
  Assess the feasibility of systematic screening for depression and anxiety using the Hospital Anxiety and Depression Scale in adult patients who are allogeneic HSCT candidates.

SECONDARY OUTCOMES:
Satisfaction among patients and providers participating in the collaborative care model | Day 0
  Assess the feasibility of implementing a collaborative care model through assessment of intervention satisfaction scores among participating patients and their health care providers.
Severity of post-transplant outcomes as defined by an investigator-designed post-transplant outcome index in relation to Hospital Anxiety and Depression Scale scores | Day 0
  Explore an association between an investigator-designed post-transplant outcome index (listed below) in patients undergoing allogeneic transplantation and Hospital Anxiety and Depression Scale scores. Aggregated outcomes abstracted from the medical record included: (a) number of days spent in hospital during transplant admission, (b) number of missed clinic appointments, (c) development of acute GVHD, (d) development of chronic GVHD, (e) admission to ICU within first 100 days of transplant, (f) date of neutrophil engraftment, (g) frequency of viral reactivation requiring antiviral treatment, and (h) death in the first 100 days.
Change in anxiety or depression as measured by the Hospital Anxiety and Depression Scale. | Day 0
  Explore whether patient's symptoms of depression and/or anxiety change over time within a collaborative care model.

CONTACTS AND LOCATIONS:
Overall Officials: Eliza M Park, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- Eliza Park, MD, Chapel Hill, North Carolina, United States